CLINICAL TRIAL: NCT01663194
Title: Observational Study of N/L Ratio in Patients With STEMI
Brief Title: Neutrophil/Lymphocyte (N/L) Ratio and Long Term Follow-up in ST-elevation Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Mahmut Akpek, Medical doctor of cardiology department, TC Erciyes University
Other Study IDs: mgkaya-makpek
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: ST Elevated Myocardial Infarction
Keywords: N/L ratio, STEMI, primary PCI, Long-term mortality
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma of blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- N/L ratio tertile 2: patients were divided in to the tertiles
  Interventions: Procedure: primary percutaneous coronary intervention, each groups
- N/L ratio tertile 3: patients were divided in to the tertiles
  Interventions: Procedure: primary percutaneous coronary intervention, each groups
- N/L ratio tertile 1: patients were divided in to the tertiles
  Interventions: Procedure: primary percutaneous coronary intervention, each groups

INTERVENTIONS:
Procedure: primary percutaneous coronary intervention, each groups — All primary PCI procedures were performed using the standard femoral approach with a 7-French guiding catheter for each patients. After administration of 5,000 IU of intravenous heparin (70 U/Kg) and a 300 mg loading dose of clopidogrel, direct stenting was performed whenever possible, and in the remaining cases, balloon pre-dilatation was performed. The operator determined the choice of stents (bare metal or drug-eluting stent).

SUMMARY:
Although the pre-procedural neutrophil to lymphocyte ratio (N/L) has been associated with adverse outcomes among patients with coronary artery disease, its role during the acute phase of ST-segment elevation myocardial infarction (STEMI) has not been fully investigated. This study sought to investigate the association of the pre-procedural N/L ratio within-hospital and long-term outcomes among STEMI patients undergoing primary percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Inflammation plays a role in the initiation and progression of the atherosclerotic process. Due to a growing recognition of its role, recent studies have focused on inflammatory markers and their association with outcomes in patients with ST-segment elevation myocardial infarction (STEMI). Recently, our single center study demonstrated that preprocedural neutrophil/lymphocyte (N/L) ratio is an independent predictor of impaired coronary flow after primary percutaneous coronary intervention (PCI) and of in-hospital major advanced cardiac events (MACE) in patients with STEMI.Several previous studies also evaluated the role of N/L ratio in long-term outcomes among patients with STEMI; however, they evaluated the association between long-term mortality and in-hospital N/L ratio, they were single-center studies and they evaluated a relatively small study population.

In the present multicenter experience, the investigators aimed to investigate the association of the preprocedural N/L ratio with the in-hospital and long-term outcomes in patients with STEMI undergoing primary PCI.

ELIGIBILITY:
Inclusion Criteria:

ST elevated myocardial infarction

Exclusion Criteria:

Treatment with fibrinolytic drugs in the previous 24 hours Active infection Previously documented history of a systemic inflammatory process Known malignancy End-stage liver disease Renal failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI patients who were admitted within 6 hours from symptom onset and who underwent primary PCI were prospectively included in this study
Sampling Method: Non-Probability Sample
Enrollment: 1034 (Actual)
Dates: Start 2000-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Akpek, MD, Study Director — Erciyes University school of medicine
Locations (1):
- Erciyes University school of medicine, Kayseri, Turkey (Türkiye)